CLINICAL TRIAL: NCT05642039
Title: Effectiveness of Mindfulness Training on the Quality of Life of Hidradenitis Suppurativa Patients
Brief Title: Mindfulness Training Hidradenitis Suppurativa (HS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hadar Lev-Tov, Associate Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20220907
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Hidradenitis Suppurativa; Quality of Life
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Course Group (Experimental): Participants will participate in the mindfulness course that would last 6 weeks.
  Interventions: Behavioral: Mindfulness Course
- HS Educational Course Group (Experimental): Participants will participate in the mindfulness course that would last 6 weeks.
  Interventions: Behavioral: HS Educational Course

INTERVENTIONS:
Behavioral: Mindfulness Course — Participants will attend a weekly 1.5-hour class over a 6-week period via Zoom. Participants will also be required to listen to guided practice audio recordings that are 12-20 minutes long and complete a weekly homework log detailing all audio recordings completed.
  Arms: Mindfulness Course Group
Behavioral: HS Educational Course — Participants will meet for 10 -15 minutes once a week over a 6-week period. The course will be administered verbally or with the use of PowerPoint slides.
  Arms: HS Educational Course Group

SUMMARY:
The purpose of this research is to investigate the effectiveness of mindfulness training on the quality of life of Hidradenitis Suppurativa (HS) patients. HS can have a profound impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Hidradenitis Suppurativa patients registered in the University of Miami Hospital dermatology system. Patients can have lesions present at the time of study participation

Exclusion Criteria:

* Individuals with any of the following: active drug addictions, untreated Post Traumatic Stress Disorder (PTSD), psychosis or suicidal ideations
* Adults unable to consent
* Pregnant women
* Prisoners
* Individuals below the age of 18 years old
* Individuals who do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
HS Quality of Life Measure (HiSQOL) Scores | Up to 10 weeks
  HS quality of life (HiSQOL) has a total score ranging from 0 to 68, with higher scores indicating more severe impact on participant's quality of life

SECONDARY OUTCOMES:
Dermatology Life Quality Index (DLQI) Scores | Up to 10 weeks
  Dermatology Life Quality Index (DLQI) has a total score ranging from 0 to 30 with the lower score indicating higher health related quality of life
Number of participants at each Refined Hurley Classification | Up to 10 weeks
  The Hurley Classification is staged as: 1 (single or multiple abscesses without sinus tract formation or scarring); 2 (recurrent abscesses with one or more sinus tracts and scarring widely separated by normal skin); 3 (diffuse involvement with multiple sinus tracts and no intervening normal skin).
Hidradenitis Suppurativa Physician's Global Assessment Scale (HS-PGA) Scores | Up to 10 weeks
  HS Physician's Global Assessment (HS-PGA) Scale is a 6-point Likert scale from 0 (clear) to 5 (very severe). Total score ranges from 0 to 30 with the higher score indicating more severe HS symptoms
Five-Facet Mindfulness Questionnaire - Short Form (FFMQ-SF) Scores | Up to 10 weeks
  FFMQ-SF has total scores ranging from 15 to 75. Higher scores indicate greater levels of mindfulness.
Pain Visual Analog Scale (VAS) Scores | Up to 10 weeks
  Pain VAS has a range from 0 to 10 with a higher score indicating worse pain
Sleep Quality Scale (SQS) Scores | Up to 10 weeks
  Sleep Quality Scale (SQS) has a score ranging from 0-10 with a greater score indicating greater sleep quality
Number of Pain medication Usage | Up to 10 weeks
  Patient reported number of pain medications used by participants in the past week
Number of work/school days missed | Up to 10 weeks
  Patient reported number of work/school days missed in the past week
Number of visits to the emergency room | Up to 10 weeks
  Patient reported number of visits to the emergency room in the past week

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Lev-Tov, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No